CLINICAL TRIAL: NCT02437916
Title: A Phase 1 First-in-Human Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 228 in Subjects With Selected Advanced Solid Tumors
Brief Title: Safety Study of AMG 228 to Treat Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140131
Record Dates: First submitted 2015-04-03; First posted 2015-05-08 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Advanced Malignancy; Advanced Solid Tumors; Cancer; Oncology; Oncology Patients; Tumors; Melanoma; Non-small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck; Transitional Cell Carinoma of Bladder; Colorectal Cancer
Keywords: Melanoma; Non-small Cell Lung Cancer (NSCLC); Squamous Cell Carcinoma; Carcinoma; Head and Neck; Transitional Cell Carinoma (TCC); Bladder; Colorectal; Colorectal Cancer (CRC)
MeSH Terms: conditions — Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Carcinoma, Squamous Cell; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMG 228 monotherapy (Experimental): Part 1 and Part 2 of the study will both be with single agent AMG 228 in different selected tumor types.
  Interventions: Drug: AMG 228

INTERVENTIONS:
Drug: AMG 228 — AMG 228 will be administered intravenously

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, anti-tumor activity, and identify a tolerable dose of AMG 228 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a pathologically documented, definitively diagnosed, advanced solid tumor
* Adequate hematological, renal, hepatic, and coagulation laboratory assessments

Exclusion Criteria:

* Active autoimmune disease, history of autoimmune disease
* Treatment with immune modulators including
* Use of warfarin, factor Xa inhibitors, or direct thrombin inhibitors
* Anti-tumor therapy (chemotherapy, antibody therapy, molecular targeted therapy, or investigational agent) within 28 days
* Major surgery within 28 days of study day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
Subject incidence of dose limiting toxicities (DLT) | 9 months
Subject incidence of treatment-emergent adverse events | 9 months
Subject incidence of treatment-related adverse events | 9 months
Subject incidence of clinically significant changes in vital signs and physical assessments | 9 months
Subject incidence of clinically significant changes in ECGs | 9 months
Subject incidence of clinically significant changes in clinical laboratory tests | 9 months
AMG 228 maximum observed concentration (Cmax) | 9 months
AMG 228 minimum observed concentration (Cmin) | 9 months
AMG 228 area under the concentration-time curve (AUC) | 9 months
AMG 228 half-life (t1/2) | 9 months

SECONDARY OUTCOMES:
Subject objective response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | 9 months
Incidence of anti-AMG 228 antibody formation | 9 months
Activation status and changes in numbers of T regulator cells (Treg) | 9 months
Subject objective response per immune-related Response Criteria (irRC) | 9 months
Activation status of cytotoxic T lymphocytes (CTL) | 9 months
Changes in numbers of cytotoxic T lymphocytes (CTL) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (3):
  - Research Site, La Jolla, California
  - Research Site, New Haven, Connecticut
  - Research Site, New York, New York
- Research Site, Parkville, Victoria, Australia
- Research Site, Leuven, Belgium
- Research Site, Villejuif, France
- Research Site, Heidelberg, Germany

REFERENCES:
- [Background] Tran B, Carvajal RD, Marabelle A, Patel SP, LoRusso PM, Rasmussen E, Juan G, Upreti VV, Beers C, Ngarmchamnanrith G, Schoffski P. Dose escalation results from a first-in-human, phase 1 study of glucocorticoid-induced TNF receptor-related protein agonist AMG 228 in patients with advanced solid tumors. J Immunother Cancer. 2018 Sep 25;6(1):93. doi: 10.1186/s40425-018-0407-x. PMID 30253804
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com